CLINICAL TRIAL: NCT04245878
Title: Interest of a Period of Fasting Before Extubation in Resuscitation Patients: a Prospective Observational Study
Brief Title: Interest of a Period of Fasting Before Extubation in Resuscitation Patients
Acronym: NUTRIGUS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: NGUYEN 2019-2
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Extubation; Intensive Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intensive care unit inpatient: Inpatient intubated resuscitation patient with a scheduled extubation
  Interventions: Other: gastric ultrasound

INTERVENTIONS:
Other: gastric ultrasound — gastric ultrasound for measurement of the antral area

SUMMARY:
Orotracheal extubation in resuscitation is a situation in which there is an elevated risk of inhalation. In resuscitation, enteral nutrition that is administered in a continuous flow is likely to accumulate in the stomach. Gastric motility in resuscitation patients may be impaired for many reasons:

* Iatrogenic: Catecholamines, sedatives and opioids slow down the digestive system and decrease the tone of the lower esophageal sphincter
* Shock, polytrauma, sepsis, pain or discomfort, or mechanical ventilation again create an alteration in gastric emptying.

Enteral nutrition is commonly discontinued to manage extubation, but it is not systematic. Discontinuation leads to a decrease in caloric intake.

Gastric ultrasound is a minimally invasive, reliable and promising means of monitoring that allows the stomach to be visualized directly. Studies on healthy subjects and in anaesthesia have made it possible to validate ultrasound in the context of the study of gastric content using both quantitative (including measurement of the antral area) and qualitative criteria. Measurement of the antral area was also studied in resuscitation. Antral area and gastric volume are closely related, with a correlation coefficient ranging from 0.6 to 0.91.

Identifying patients at risk of inhalation by ultrasound could allow individualized enteral nutrition management prior to extubation in the resuscitation unit, and thus optimize nutritional management.

The objective of the study is to identify factors associated with greated antral area in patients hospitalized in the intensive care unit. The hypothesis is that continued enteral nutrition before extubation is associated with increased gastric volume as measured by ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Person or next of kin/designated representative has provided his or her non-opposition
* Patient in medical or surgical intensive care, admitted for an urgent medical or surgical reason and for whom extubation have been planned by the practitioner in charge of the patient

Exclusion Criteria:

* Person subject to legal protection (guardianship, trusteeship)
* Person subject to a justice safeguard measure
* Pregnant, parturient or breastfeeding woman
* Minor
* Anechoic patient or patient without an exploitable ultrasound window
* History of gastric or esophageal surgery
* Limitation of Care (LOC) order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care patients receiving respiratory assistance by mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Surface of the antral area in mm² | pre-extubation
Duration of enteral feeding interruption in hours | pre-extubation

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Nguyen M, Drihem A, Berthoud V, Dransart-Raye O, Bartamian L, Gounot I, Guinot PG, Bouhemad B. Fasting does not guarantee empty stomach in the intensive care unit: A prospective ultrasonographic evaluation (The NUTRIGUS study). Anaesth Crit Care Pain Med. 2021 Dec;40(6):100975. doi: 10.1016/j.accpm.2021.100975. Epub 2021 Nov 4. PMID 34743035